CLINICAL TRIAL: NCT04994743
Title: Multiple Dose Safety, Tolerability, Plasma and Cerebrospinal-Fluid Pharmacokinetic Study of Oral Doses of CORT113176
Brief Title: Safety, Tolerability, and Pharmacokinetic Study of CORT113176 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Corcept Therapeutics (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: CORT113176-653; 2021-002456-36 (EudraCT Number)
Record Dates: First submitted 2021-07-29; First posted 2021-08-06 (Actual); Last update posted 2021-10-11 (Actual); Status verified 2021-10

CONDITIONS: Healthy Adults
MeSH Terms: interventions — CORT113176

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- Cohort 1: CORT113176 150 mg (Experimental): Participants will receive CORT113176 150 mg lipid capsule formulation by mouth once daily under fed conditions for 14 days.
  Interventions: Drug: CORT113176
- Cohort 1: Placebo matching CORT113176 (Placebo Comparator): Participants will receive placebo matching CORT113176 capsule by mouth once daily under fed conditions for 14 days.
  Interventions: Drug: Placebo matching CORT113176
- Cohort 2: CORT113176 300 mg (Experimental): Participants will receive CORT113176 300 mg lipid capsule formulation by mouth once daily under fed conditions for 14 days. Progression from Cohort 1 to 2 will be done based on safety and tolerability outcome from Cohort 1 and only after Cohort 1 has received study drug for ≥7 days.
  Interventions: Drug: CORT113176
- Cohort 2: Placebo matching CORT113176 (Placebo Comparator): Participants will receive placebo matching CORT113176 capsule by mouth once daily under fed conditions for 14 days.
  Interventions: Drug: Placebo matching CORT113176
- Cohort 3: CORT113176 ≥300 mg (Experimental): Participants will receive CORT113176 ≥300 mg not to exceed 450 mg lipid capsule formulation by mouth once daily under fed conditions for 14 days. Cohort 3 is optional, and progression from Cohort 2 to 3 be done based on safety and tolerability outcome from Cohort 2 and only after Cohort 2 has received study drug for ≥7 days.
  Interventions: Drug: CORT113176
- Cohort 3: Placebo matching CORT113176 (Placebo Comparator): Participants will receive placebo matching CORT113176 capsule by mouth once daily under fed conditions for 14 days.
  Interventions: Drug: Placebo matching CORT113176

INTERVENTIONS:
Drug: CORT113176 — CORT113176 lipid capsule formulation for oral administration
  Arms: Cohort 1: CORT113176 150 mg; Cohort 2: CORT113176 300 mg; Cohort 3: CORT113176 ≥300 mg
Drug: Placebo matching CORT113176 — Placebo matching CORT113176 lipid capsule formulation for oral administration
  Arms: Cohort 1: Placebo matching CORT113176; Cohort 2: Placebo matching CORT113176; Cohort 3: Placebo matching CORT113176

SUMMARY:
This is a safety, tolerability, and pharmacokinetic study in 2 cohorts of healthy male participants with an option for an additional cohort. Cohorts 1 and 2 will receive once daily by mouth CORT113176 150 mg and 300 mg, respectively, for 14 days under fed conditions. Progression from Cohort 1 to Cohort 2 will be done based on the safety and tolerability outcome in Cohort 1 and after Cohort 1 has received the study drug for at least 7 days. The optional Cohort 3 may receive a higher dose that will not exceed CORT113176 450 mg once daily by mouth for 14 days under fed conditions. The progression from Cohort 2 to the optional cohort (Cohort 3) will be based on the same precautions as with the progression from Cohort 1 to Cohort 2. Each participant will undergo safety evaluations. Pharmacokinetics of CORT113176 will be assessed in plasma and cerebrospinal fluid (CSF) samples. Pharmacodynamic assessments will include the measurement of serum cortisol.

ELIGIBILITY:
Inclusion Criteria:

* Body mass index (BMI) of 18.0 to 30.0 kg/m^2, inclusive
* Body weight ≤100 kg.
* Must agree to adhere to the requirements on contraception, exposure to sexual partners, and sperm donation as defined in the protocol
* Additional criteria apply.

Exclusion Criteria:

* Received any investigational drug in a clinical research study within the last 90 days
* History of alcohol abuse or drug addiction (including soft drugs like cannabis products) within past 5 years.
* Regular alcohol consumption
* Positive drug, nicotine (cotinine), or alcohol screen
* Current smokers, user of e-cigarettes and nicotine replacement products and those who have used these products within the last 3 months
* Have a pregnant partner
* Clinically significant abnormal clinical chemistry, hematology (including coagulation), or urinalysis
* Positive hepatitis B surface antigen (HBsAg), hepatitis C virus (HCV) antibody or human immunodeficiency virus (HIV) results
* Positive nasopharyngeal polymerase chain reaction (PCR) test for severe acute respiratory syndrome Covid Virus-2 (SARS-CoV-2) on Day -1 or within 8 weeks prior to screening.
* Contact with COVID-19 positive (or suspected) persons within 14 days prior to first dose
* Active renal and/or hepatic disease
* History of clinically significant cardiovascular, renal, hepatic, endocrine, metabolic, respiratory, gastrointestinal (GI), neurological, or psychiatric disorder
* Abnormalities in brain and lumbar spine, or other medical or surgical conditions or clinically significant abnormal findings, for which lumbar puncture is contraindicated
* History of clinically significant back pain, back pathology and/or back injury
* History of significant active bleeding or coagulation disorder or have taken non-steroidal anti-inflammatory drugs or other drugs that affect coagulation or platelet function within 14 days prior to lumbar puncture
* Allergy to lidocaine (Xylocaine®) or its derivatives
* Any form of cancer within the 5 years (exceptions apply)
* History and/or symptoms of adrenal insufficiency
* Have a condition that could be aggravated by glucocorticoid antagonism
* Donation or loss of greater than 400 mL of blood within the previous 3 months
* Currently using glucocorticoids or have a history of systemic glucocorticoid use at any dose within the last 12 months or 3 months for inhaled products
* Additional criteria apply.

Ages: 18 Years to 65 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 16 (Actual)
Dates: Start 2021-07-13 (Actual); Primary Completion 2021-09-30 (Actual); Study Completion 2021-09-30 (Actual)

PRIMARY OUTCOMES:
Number of Participants with One or More Adverse Events | Up to Day 28

SECONDARY OUTCOMES:
Maximum Plasma Concentration (Cmax) of CORT113176 | Before dosing and a pre-specified time points up to Day 17
Time of Cmax (Tmax) of Plasma CORT113176 | Before dosing and a pre-specified time points up to Day 17
Apparent Elimination Half-life (t1/2) of Plasma CORT113176 | Before dosing and a pre-specified time points up to Day 17
Area Under the Plasma Concentration-time Curve (AUC) of Plasma CORT113176 | Before dosing and a pre-specified time points up to Day 17
Cerebrospinal Fluid Concentration of CORT113176 | Approximately 3 and 5 hours after dosing on Day 7
Serum Concentration of Cortisol | Before and approximately 12 hours after dosing on Days 1, 7, and 14

CONTACTS AND LOCATIONS:
Overall Officials: Hazel Hunt, Ph.D., Study Director — Corcept Therapeutics
Locations (1):
- Site 01, Groningen, Netherlands

IPD SHARING:
Plan to Share IPD: No